CLINICAL TRIAL: NCT06181279
Title: Effects of Individualized Positive End-expiratory Pressure Guided by Driving Pressure on Postoperative Atelectasis After Bariatric Surgery in Patients With Morbid Obesity: A Single-center, Prospective, Randomized Controlled Study
Brief Title: Effects of Individualized PEEP Guided by Driving Pressure on Postoperative Atelectasis in Patients With Morbid Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yongtao Sun (Other)
Responsible Party: Sponsor-Investigator, Yongtao Sun, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DP guided PEEP
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Atelectasis; Obesity, Morbid
Keywords: Individual Positive End-expiratory Pressure; Driving Pressure; Ventilator-induced Lung Injury
MeSH Terms: conditions — Pulmonary Atelectasis; Obesity, Morbid; Ventilator-Induced Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized PEEP group (Experimental): After recruitment maneuver, PEEP is titrated decreasingly using driving pressure guided individualised PEEP ventilation strategy, and the PEEP corresponding to the lowest driving pressure is the individualised PEEP.
  Interventions: Procedure: Individualized PEEP group
- Fixed PEEP group (Other): After recruitment maneuver, PEEP is fixed at 8cmH2O.
  Interventions: Procedure: Fixed PEEP group

INTERVENTIONS:
Procedure: Individualized PEEP group — Individualized PEEP group: Recruitment Maneuver (RM) is performed first. In pressure control mode, PEEP and airway plateau pressure are increased to 20 cmH2O and 35 cmH2O at a rate of 5 cmH2O every 30s, and driving pressure is maintained at 15 cmH2O throughout. Subsequently, in volume-controlled ventilation mode, PEEP decreases from 20 cmH2O to 4 cmH2O at gradient of 2 cmH2O, and each PEEP level is maintained for 30s. The PEEP corresponding to the lowest driving pressure is the individualized PEEP we need. If multiple PEEP levels showed the same lowest driving pressure, the lowest PEEP value as the individualized PEEP. The above procedures are performed three times during the surgery (5 minutes after intubation,5 minutes after the beginning of pneumoperitoneum, and 5 minutes after the end of pneumoperitoneum).
  Arms: Individualized PEEP group
Procedure: Fixed PEEP group — After the same RM, PEEP is fixed at 8 cmH2O.
  Arms: Fixed PEEP group

SUMMARY:
Atelectasis is a common complication in patients undergoing surgery under general anesthesia, particularly in obese patients. Postoperative atelectasis could last for more than 24h and contribute to a variety of other complications, including hypoxemia and pneumonia. We plan to conduct a single-center, randomized controlled trial in patients undergoing bariatric surgery to test the hypothesis that driving pressure guided PEEP could reduce the postoperative atelectasis.

DETAILED DESCRIPTION:
Positive end-expiratory pressure (PEEP) is a strategy that helps to keep alveoli open during surgery and to prevent postoperative atelectasis. A fixed PEEP without considering the respiratory mechanics in individual patients, however, is not optimal. Individualized PEEP therefore has been increasingly studied, and has been shown to improve oxygenation in both nonobese and obese patients. Studies have shown that the occurrence and prognosis of PPCs are significantly associated with high driving pressure (DP), but not with VT and PEEP. Driving pressure-guided individualized PEEP is expected to be a novel perioperative lung protection strategy. Consequently, the main aim of this study is to investigate the effect of a driving pressure-guided individualized PEEP ventilation strategy on postoperative pulmonary atelectasis in morbidly obese patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years old;
* Body mass index (BMI) ≥ 40 kg/m2;
* ASA classification I to III;
* Signing the informed consent form for this clinical study;

Exclusion Criteria:

* Respiratory infection within 4 weeks; severe respiratory system diseases; history of pulmonary and/or thoracic surgery; neuromuscular dysfunction;
* Serious cardiac, renal or haematopoietic diseases;
* Contraindications to PEEP；

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary atelectasis | After 30 minutes of extubation
  The primary outcome of this study is postoperative atelectasis measured by lung ultrasound. Each hemithorax is divided into 6 regions using 3 longitudinal lines (parasternal, anterior and posterior axillary)and 2 axial lines (one above the diaphragm and the other 1 cm above the nipples). The 12 lung regions were scanned sequentially from right to left, cranial to caudal and anterior to posterior. Each region is assessed using a 2-dimen-sional view with the probe placed parallel to the ribs. It distinguishes four progressive steps of loss of aeration according to the artifacts visualized in a scan: score 0, normal aeration (A-lines or no more than two B-lines); score 1, moderate loss of aeration (three or more well-spaced B-lines); score 2, severe loss of aeration(coalescent B-lines); and score 3, complete loss of aeration(tissue-like pattern). We define atelectasis to be significant if any region had a lung consolidation score of ≥2.

SECONDARY OUTCOMES:
Postoperative pulmonary ultrasound score | After 30 minutes of extubation
  Each hemithorax is divided into 6 regions using 3 longitudinal lines (parasternal, anterior and posterior axillary)and 2 axial lines (one above the diaphragm and the other 1 cm above the nipples). The 12 lung regions were scanned sequentially from right to left, cranial to caudal and anterior to posterior. Each region is assessed using a 2-dimen-sional view with the probe placed parallel to the ribs. It distinguishes four progressive steps of loss of aeration according to the artifacts visualized in a scan: score 0, normal aeration (A-lines or no more than two B-lines); score 1, moderate loss of aeration (three or more well-spaced B-lines); score 2, severe loss of aeration(coalescent B-lines); and score 3, complete loss of aeration(tissue-like pattern). We define atelectasis to be significant if any region had a lung consolidation score of ≥2. Based upon the LUS scoring system, each area is scored from 0-3, so a minimum zero or maximum 36 score is possible.

CONTACTS AND LOCATIONS:
Overall Officials: yong t Sun, Ph.D, Study Chair — Shandong First Medical University
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Derived] Ren Y, Sun YT, Zhang P, Chen L, Liu P, Zhou Z, Wang Y. Effect of driving pressure-guided individualised positive end-expiratory pressure on postoperative atelectasis in patients with morbid obesity: study protocol of a randomised controlled trial. BMJ Open. 2025 Mar 6;15(3):e091217. doi: 10.1136/bmjopen-2024-091217. PMID 40050061